CLINICAL TRIAL: NCT03571451
Title: A Multi-center Prospective Cohort Study Based on Peritoneal Dialysis Telemedicine-assisted Platform
Acronym: PDTAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Collaborators: The Second Hospital of Hebei Medical University (Other); Army Medical University, China (Other); The First Affiliated Hospital of Zhengzhou University (Other); Hebei Medical University Third Hospital (Other); Peking University Shenzhen Hospital (Other); Handan Central Hospital (Other); Beijing Haidian Hospital (Other); People's Hospital of Qinghai Province (Unknown); Cangzhou Central Hospital (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Shengjing Hospital (Other); The Second Hospital of Anhui Medical University (Other); Peking University People's Hospital (Other); The First Affiliated Hospital of BaoTou Medical College (Other); The People's Hospital of Chuxiong Yi Autonomous Prefecture (Unknown); Beijing miyun district hospital (Unknown); Second Hospital of Shanxi Medical University (Other); People's Hospital of Gansu (Unknown); Pingdingshan first people's Hospital (Unknown); The first people's hospital of Xining (Unknown); The First Hospital of Jilin University (Other); Cangzhou People's Hospital (Other); Taiyuan central hospital (Unknown); People's hospital of Langfang (Unknown); China Rehabilitation Research Center (Other Government); Dongzhimen Hospital, Beijing (Other); Department of Epidemiology and Biostatistics, School of Public Health, Peking University (Unknown); Department of Statistics, Peking University First Hospital (Unknown)
Responsible Party: Principal Investigator, Dong Jie, Director of Peritoneal dialysis center, Peking University First Hospital
Other Study IDs: PDTAP study
Record Dates: First submitted 2018-06-20; First posted 2018-06-27 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Peritoneal Dialysis
Keywords: peritoneal dialysis; survival rate; technique survival rate; risk factors; end stage renal disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All participants were voluntary to collect the blood, urine, DNA and tissue specimen and signed the informed consent form.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Increasing the proportion of patients on peritoneal dialysis (PD) may relieve the financial burden caused by the growing number of patients with end-stage renal disease (ESRD). The investigators are developing a PD database in China using peritoneal dialysis telemedicine-assisted platform (PD TAP). The survival rate and technique survival rate of PD patients, as well as risk factors associated with survival and technique survival will be analyzed through PD TAP.

DETAILED DESCRIPTION:
The growing number of patients with ESRD leads to an increasing medical burden all around the world. Patients on PD have a similar long-term survival rate as patients on hemodialysis, with a much lower cost of medical resources. Therefore, increasing the percentage of patients on PD may relieve the increasing financial burden for the whole society.

Of note, technique survival and patient survival in PD still need to be improved. Based on results from multi-center cohort studies, some prognostic factors have been explored and intervened in recent years. However, robust data from large samples on potential predictors pertaining to patients' clinical characteristics, and PD practice on clinical outcomes in the real world is still limited. This phenomenon calls an action on exploring novel risk factors of patient outcome, especially through national-level prospective cohort study.

The investigators are developing a national-level PD database by registering all patients receiving PD on PD TAP. The study is underway in 27 hospitals from 14 provinces located at 7 geographical regions (northwest, northeast, north, central, southwest, southeast and south) in China. National samples of PD units are recruited based on the availability of professional PD team who is willing participant and could regularly follow participants. Our study aims to enroll adult 7,000 patients with end stage renal disease receiving PD. Patients-, treatment- and telemedicine-level variables are collected at baseline and thus at 3-month intervals. PD practice surveys are collected at baseline. All-cause mortality and transfer to hemodialysis will be recorded as primary outcomes. Other clinical outcomes including infectious and non-infectious complications would be recorded. Apart from the above objectives, potential collaboration between PDTAP and local or international clinical research could develop ancillary studies with specific aims. Examples of key research and ancillary investigation proposed in PDTAP study are as follows: 1) Long-term effects of telemedicine on clinical outcomes of patients on PD: a propensity matched study, 2) Anemia, erythrocyte-stimulating agents, inflammation and the association with mortality in patients on PD, 3) The management of serum calcium, phosphate, and hyperparathyroidism and its relationship with mortality in patients on PD, 4) The prevalence of hypomagnesemia, and all-cause and cardiovascular mortality in patients on PD, 5) The prevalence, predictors, and outcomes of PD-related peritonitis, 6) Association between hemoglobin levels and serum albumin levels and mortality in diabetic and non-diabetic patients on PD, 7) Glucose absorption (measured as the difference between the amount of glucose in peritoneal dialysate absorbed into the peritoneal cavity in 24h and that measured in the 24h drained effluent) and its association with metabolic syndrome, cardiovascular events, and mortality in patients on PD. The follow-up will be continued until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal disease patients receiving maintenance peritoneal dialysis;
* more than 14 years old

Exclusion Criteria:

* receiving temporary PD due to acute kidney injury
* loss to follow up without any outcomes recorded.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with end-stage renal disease receiving maintenance peritoneal dialysis
Sampling Method: Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
All-cause death | 10 years
  All-cause death refers to the number of patients who died within the anticipated time frame. For example death caused by CVD, systemic infection, malignancies (according to the WHO classification), and protein-energy wasting.
Transfer to hemodialysis | 10 years
  Transfer to hemodialysis refers to the number of patients who were Transfer to hemodialysis from PD due to any cause within the anticipated time frame. For example, caused by dialysis inadequacy, volume overload, infection-related (peritonitis and exitsite infection), catheter dysfunction (catheter blockage and displacement), ultrafiltration failure, et al.

SECONDARY OUTCOMES:
Peritonitis | 10 years
  The incidence of peritoneal dialysis related peritonitis during the time frame. Includes first-episode/multi-episode, refractory, relapsing, repeat, and recurrent, organism-specific, peritonitis-related death or transfer to hemodialysis.
Exit-site/tunnel infection | 10 years
  The incidence of exit-site/tunnel infection during the time frame. Includes organism-specific, infection-related death or transfer to hemodialysis.
Cardiovascular events | 10 years
  The incidence of cardiovascular events during the time frame. For example, caused by congestive heart failure, angina or acute myocardial infarction, cerebrovascular accident, and peripheral arterial events.
Abdominal wall complications | 10 years
  The incidence of abdominal wall complications occurred during the time frame, such as peritoneal leaks and hernia.
others | 10 years
  The incidence of other complications during the time frame, such as new-onset diabetes/cancer, and encapsulating peritoneal sclerosis.
Other causes for terminating PD | 10 years
  The incidence of other causes for terminating PD during the time frame. For example, caused by kidney transplantation, burnout, caretaker burnout or absence physical handicap preventing self-care.

CONTACTS AND LOCATIONS:
Locations (27):
- China (27):
  - The second affiliated hospital of Anhui Medical University, Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - People's Hospital of Gansu Province, Lanzhou, Gansu
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Cangzhou central hospital, Cangzhou, Hebei
  - People's hospital of Cangzhou, Cangzhou, Hebei
  - Handan Central Hospital, Handan, Hebei
  - People's hospital of Langfang, Langfang, Hebei
  - The second hospital of Hebei medical university, Shijiazhuang, Hebei
  - The third hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The second affiliated hospital of Harbin Medical University, Harbin, Heilongjiang
  - Pingdingshan People's Hospital No.1, Pingdingshan, Henan
  - First affiliated hospital of Zhengzhou University, Zhengzhou, Henan
  - The first affiliated hospital of Baotou Medical College, Baotou, Inner Mongolia
  - The first hospital of Jilin University, Changchun, Jilin
  - Shengjing hospital affiliated to China Medical University, Liaoyang, Liaoning
  - People's Hospitel of Qinghai Province, Xining, Qinghai
  - The first people's hospital of Xining, Xining, Qinghai
  - Taiyuan central hospital, Taiyuan, Shanxi
  - The second hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The People's Hospital of Chuxiong Yi Autonomous Prefecture, Chuxiong, Yunnan
  - Beijing Charity Hospital, Beijing
  - Beijing dongzhimen Hospital, Beijing
  - Beijing haidian hospital, Beijing
  - Beijing miyun district hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Xinqiao hospital of the Third Military Medical University, Chongqing

REFERENCES:
- [Derived] Li X, Ma T, Hao J, Song D, Wang H, Liu T, Xu X, Dong J. The relationship between exercise and the occurrence of abdominal wall complications in patients on peritoneal dialysis. BMC Nephrol. 2025 Jul 15;26(1):389. doi: 10.1186/s12882-025-04317-7. PMID 40665238